CLINICAL TRIAL: NCT06233682
Title: The Enriched Environment as an Integrated Tool in the Ward Setting for Improving Functional Outcome in People With Acute Stroke: a Study Within the Neurological Clinic Unit
Brief Title: The Enriched Environment as an Integrated Tool in the Ward Setting
Acronym: ENVIRONMENT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Alessandra Del Felice, Associate Professor of Physical and Rehabilitation Medicine, University of Padova
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PROTOCOL_ENVIRONMENT
Record Dates: First submitted 2023-11-27; First posted 2024-01-31 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Stroke; Stroke, Acute
Keywords: enriched environment; in-patients setting
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Longitudinal interventional study in which participants are not randomised, as the experimental design alternates sequentially between the control and experimental groups, with no possibility of interaction between the two groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enriched environment group (Experimental): 25 people with stroke recruited from the acute in-patient ward of the Neurology Clinic, meeting the inclusion criteria.
  Interventions: Other: Enriched environment
- No intervention (No Intervention): 25 people with stroke recruited from the acute in-patient ward of the Neurology Clinic, meeting the inclusion criteria.

INTERVENTIONS:
Other: Enriched environment — In the experimental group (enriched environment), assistants will supervise participants sponatneoulsy engaging in activities, including listening to music, drawing, playing cards or board games, exercising the affected upper limb with constructions or puzzles, etc., in the living room and personal rooms. Posters and clocks will also aid in orientation and improve the physical environment.
  Arms: Enriched environment group

SUMMARY:
The goal of this longitudinal interventional study is to integrate the enriched environment (EE) in the context of the Neurology Clinic ward of the General Hospital - University of Padua, by verifying its effectiveness and impact on psychological well-being, functional recovery, activity level, and quality of life in people with stroke.

DETAILED DESCRIPTION:
The EE will be integrated within the shared areas of the Neurology ward and in inpatient rooms, providing materials and aids to encourage physical, cognitive and social activity. The study will recruit for 9 months plus 6 months of follow-up. It will recruited a total of 50 people with stroke (25 for experimental and control group). After providing informed consent, participants will be evaluated on admission, at discharge, at 4 weeks (follow-up phone interview) and at 6 months (telephone interview). Participants will be psuedo randomized, as the ward will be environmentally enriched during consecutive alternating time frames. The instrument used to measure the multidimensional recovery will be the Stroke Impact Scale. Specific secondary outcomes will assessed the recovery in motor, cognitive and communication function, the impact on physical activity, mood, the type of activity of participants exposed to EE and the impact on the ward organization.

ELIGIBILITY:
Inclusion Criteria:

* Ischaemic or haemorrhagic stroke, in any territory, occurring at least 24 hours before enrollment;
* Participant consent to participate in the study;
* Mecial stabilisation.

Exclusion Criteria:

* Uncooperative participant, as assessed by theMontreal Cognitive Assessment scale < 15
* medically not stabtability and/or reduced level of consciousness and/or psychomotor agitation;
* Lack of trunk control (score <12 in item 3 of the Trunk Control Test: balance in sitting position) such that it is impossible to maintain a sitting position or a safe posture in a wheelchair;
* Speech evaluation confirming comprehension aphasia hampering understanding of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Stroke Impact Scale | T0: baseline (enrollment), T1: immediately after intervention (discharge), T2: 4 weeks post intervention (telephone interview), T3: 6 months post intervention (telephone interview)
  The Stroke Impact Scale (SIS) is a self-report questionnaire that evaluates disability and health-related quality of life after stroke. SIS is a 59-item measure. Each item is rated in a 5-point Likert scale in terms of the difficulty the patient has experienced in completing each item. Summative scores are generated for each domain, scores range from 0-100.

SECONDARY OUTCOMES:
Functional Independence Measure (FIM) scale | T0: baseline (enrollment), T1: immediately after intervention (discharge), T2: 4 weeks post intervention (telephone interview), T3: 6 months post intervention (telephone interview)
  Functional Independence Measure (FIM) scale is used to assess and grade the functional status of a person based on the level of assistance he or she requires. FIM is comprised of 18 items, grouped into 2 subscales - motor and cognition. Each item is scored on a 7 point ordinal scale, ranging from a score of 1 to a score of 7. The higher the score, the more independent the patient is in performing the task associated with that item. The total score for the FIM instrument (the sum of the motor and cognition subscale scores) will be a value between 18 and 126.
Functional Assessment Test for Upper Limb | T0: baseline (enrollment), T1: immediately after intervention (discharge)
  The Functional Assessment Test for Upper Limb (FAST-UL) is a clinical scale based on observational movement analysis of UL impairment in stroke survivors, composed of 5 items measured through a 4-level ordinal scale.The items identified by the panel of experts are Hand to Mouth (HtM), RtT, PS, GaR, and PaR.
Functional Ambulatory Category (FAC) | T0: baseline (enrollment), T1: immediately after intervention (discharge), T2: 4 weeks post intervention (telephone interview), T3: 6 months post intervention (telephone interview)
  The Functional Ambulation Categories (FAC) is a 6-point functional walking test that evaluates ambulation ability, determining how much human support the patient requires when walking, regardless of whether or not they use a personal assistive device. Scoring range from 0: nonfunctional ambulator to 5: Ambulator, independent.
Dynamic Gait Index (DGI) if FAC > 3 | T0: baseline (enrollment), T1: immediately after intervention (discharge)
  The Dynamic Gait Index (DGI) is a clinical tool used to assess gait, balance and fall risk. It evaluates not only the usual steady-state walking, but also walking during more challenging tasks. Scores are based on a 4-point scale. Highest possible score is 24 points.
Oxford Cognitive Screening (OCS) | T0: baseline (enrollment), T1: immediately after intervention (discharge)
  The Oxford Cognitive Screen (OCS) is a first-line, stroke-specific and domain-specific cognitive screening tool which can be delivered at the bedside in acute stroke.
Typical values of Physical Activity Level (PAL) | T0: baseline (enrollment), T1: immediately after intervention (discharge), T2: 4 weeks post intervention (telephone interview), T3: 6 months post intervention (telephone interview)
  The physical activity level (PAL) is a way to express a person's daily physical activity as a number, and is used to estimate a person's total energy expenditure. Ranges: Extremely inactive PAL <1.40 - Extremely active PAL >2.40.
Hospital Anxiety and Depression Scale (HADS) | T0: baseline (enrollment), T1: immediately after intervention (discharge), T2: 4 weeks post intervention (telephone interview), T3: 6 months post intervention (telephone interview)
  Hospital Anxiety and Depression Scale (HADS) is used to determine the levels of anxiety and depression. The HADS is a fourteen item scale. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression.
Motor Activity Log | T2: 4 weeks post intervention (telephone interview), T3: 6 months post intervention (telephone interview)
  Individuals are asked to rate Quality of Movement (QOM) and Amount of Movement (AOM) during daily functional tasks.
  Target tasks include object manipulation (e.g. pen, fork, comb, and cup) as well as the use of the arm during gross motor activities (e.g. transferring to a car, steadying oneself during standing, pulling a chair into a table while sitting). Items scored on a 6-point ordinal scale.
Ad hoc behavioral mapping checklist | T0: baseline (enrollment), T1: immediately after intervention (discharge)
  Tool created to quantify and study the type of activity (physical, cognitive, social) carried out by participants.
Ad hoc questionnaire for health care workers | T1: post intervention
  Assessing impact on ward organisation.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Del Felice, MD, PhD, Principal Investigator — University of Padova
Locations (1):
- Teaching Hospital, University of Padova, Padua, Italy

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data sheet
Supporting Information: Study Protocol, CSR
Time Frame: Upon study completion
Access Criteria: Upon direct request of researchers providing any official reaserch identification (ORCID, Reaserch ID, etc)